CLINICAL TRIAL: NCT01630291
Title: A Non-Randomized, Open-Label Study to Determine the Effect of Electrical Stimulation on Tear Production
Brief Title: The Effect of Electrical Stimulation on Tear Production
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oculeve, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OCU-002
Record Dates: First submitted 2012-06-15; First posted 2012-06-28 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Electrodes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Electrical stimulation (Experimental)
  Interventions: Device: Electrode device

INTERVENTIONS:
Device: Electrode device — Lacrimal gland stimulation
  Other Names: External Neurostimulator Trialing System (Medtronic)

SUMMARY:
The purpose of this study is to investigate whether electrical stimulation of the nerve innervating the tear gland results in tear production in subjects with severe Dry Eye.

DETAILED DESCRIPTION:
A non-randomized, open-label study designed to investigate the feasibility of a novel treatment for severe Dry Eye Disease, which involves safe delivery of small electrical currents to the lacrimal nerve to induce tear production.

ELIGIBILITY:
Inclusion Criteria:

* Schirmer test with topical anesthesia of ≤ 5 mm/5 min in at least one eye
* Sum of corneal and interpalpebral conjunctival staining of > +5 in the same eye where corneal staining is > +2 using the CLEK criteria.

Exclusion Criteria:

* Individuals with the presence or history of any ocular disorder or condition (including ocular surgery, trauma, and disease) that could possibly interfere with the interpretation of the study results. Individuals who have had LASIK or other refractive surgeries are eligible. Excluded conditions include:

  * History of orbital trauma
  * History of orbital surgery
  * Orbital cancer
  * History of orbital cancer
* Within the 3 months before the Screening Visit, known history of ocular infection (viral, bacterial, fungal), inflammation not associated with dry eye, or active ocular herpes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-07; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Schirmer Score | Up to 16 days

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Salcedo, M.D., Principal Investigator — Asociación para Evitar la Ceguera en México
Locations (1):
- APEC, La Concepción, Mexico City, Mexico